CLINICAL TRIAL: NCT04607174
Title: Measuring Voluntary Activation of the Quadriceps Femoris During Isokinetic Concentric Contractions with the Interpolated Twitch Technique (ITT) in Subjects with Neuromotor Disorders
Brief Title: Voluntary Activation During Isokinetic Contractions in Subjects with Neuromotor Disorders
Acronym: ATTILA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Luigi Tesio, Prof, MD, Director of the Department of Neuromotor Rehabilitation, Ospedale San Luca, Istituto Auxologico Italiano, IRCCS; Full Professor, Department of Biomedical Sciences for Health, Università degli Studi di Milano, Milan, Italy, Istituto Auxologico Italiano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24C903
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Poststroke/CVA Hemiparesis; Parkinson Disease; Knee Impairment
Keywords: voluntary activation; lower limb; interpolated twitch technique; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pathologic group (Other): At least 20 participants with various neurologic or orthopaedic conditions (for example, hemiparesis post-stroke, multiple sclerosis, traumatic knee injuries, knee osteoarthritis) will be enrolled.
  Interventions: Other: Pathologic group

INTERVENTIONS:
Other: Pathologic group — Voluntary Activation level will be determined according to the interpolate twitch technique (ITT).
  During isometric contractions (knee at 40° flexion), three electric shocks (doublets) will be delivered. The first shock will be delivered at rest before contraction. The second one will be delivered 3-4 s after the beginning of the effort. The third one will be delivered at rest 2-3 s after the contraction has ended. Two isometric contractions will be performed, with a 3-minute break.
  Then, 3 consecutive continuous passive motion (CPM) extension-flexions of the knee joint (range 105-0°), and 3 isokinetic concentric contractions (ISOK) will be performed. During both CPM and ISOK an electric shock will be delivered during each repetition. The instant of stimulation will be determined in a way allowing the twitch moments to peak at exactly 40° of knee flexion during extension. The same procedure will be administered first to the affected limb, and then to the non-affected limb.

SUMMARY:
Activation is the amount of voluntary recruitment of a muscle during voluntary contraction. Full activation implies the recruitment of all muscle fibres at their tetanic frequency. In healthy subjects, and even in sports performances, full activation may be rarely achieved despite a subjectively maximal effort.

Highly decreased activation has been observed in patients affected by various orthopaedic and neurological disorders. In these subjects, paresis may be caused or aggravated by primitive impairments of the central nervous system and/or, by stimuli arising from peripheral damaged tissues that inhibit the corticospinal or the intraspinal recruitment of motoneurones ("arthrogenous muscle weakness"). There are numerous investigations in the literature on activation measured during isometric contractions, while they are substantially missing as far as isokinetic concentric contractions are concerned. There are reasons to suppose that, contrary to what has been demonstrated for healthy subjects, in patients with various motor impairments the activation is diminished the more, the higher is the joint rotation speed.

The present study aims to investigate the amount of activation of the quadriceps femoris during subjectively maximal isometric contractions at 40° knee flexion (0°=complete extension) and isokinetic concentric contractions at an angular velocity of 100°/s in patients with various orthopaedic and neurologic conditions.

Activation will be measured on an isokinetic dynamometer, through the "interpolated twitch technique". This consists of stimulating a representative sample of the muscle belly through an electric shock. If the shock does not generate an extra force during contraction, all muscle fibres belonging to the sample reached by the electric shock can be claimed to be recruited at their tetanic frequency. Otherwise, following the stimulus, a twitch can be observed revealing submaximal voluntary recruitment of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years old;
* ability to sign the informed consent form;
* ability to understand the instructions and to complete the motor task;
* voluntary knee flexion-extension range of at least 70°;
* maximal extension of angle < 30° (0°=full extension, 180° sagittal tibio-femural angle).

Exclusion Criteria:

* pregnancy;
* a history of epilepsy (to avoid the risk for seizures triggered by the stimuli);
* Mini Mental State Examination ≤27/30;
* implanted electro-sensitive devices;
* any orthopedic condition limiting the articular mobility or muscular strength of the lower limbs;
* current treatment with oral anticoagulant therapy (to avoid the risk for muscle hemorrhage);
* medium/serius osteoporosis (femoral Bone Mineral Density on the affected side, t-score < (-3.5));
* familiarity with the testing method.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Voluntary Activation | Day 1
  Voluntary Activation = [1 - (Interpolated Twitch/Resting Twitch)]%, where Interpolated Twitch and Resting Twitch are the peak torques caused by the electric shock during the voluntary contraction and a rest, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Tesio, MD, Full professor, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Babault N, Pousson M, Ballay Y, Van Hoecke J. Activation of human quadriceps femoris during isometric, concentric, and eccentric contractions. J Appl Physiol (1985). 2001 Dec;91(6):2628-34. doi: 10.1152/jappl.2001.91.6.2628. PMID 11717228
- [Background] Behrens M, Husmann F, Gube M, Felser S, Weippert M, Bruhn S, Zschorlich V, Mau-Moeller A. Intersession reliability of the interpolated twitch technique applied during isometric, concentric, and eccentric actions of the human knee extensor muscles. Muscle Nerve. 2017 Aug;56(2):324-327. doi: 10.1002/mus.25498. Epub 2017 Apr 12. PMID 27935064
- [Background] Behrens M, Mau-Moeller A, Mueller K, Heise S, Gube M, Beuster N, Herlyn PK, Fischer DC, Bruhn S. Plyometric training improves voluntary activation and strength during isometric, concentric and eccentric contractions. J Sci Med Sport. 2016 Feb;19(2):170-6. doi: 10.1016/j.jsams.2015.01.011. Epub 2015 Feb 4. PMID 25766509
- [Background] Beltman JG, Sargeant AJ, van Mechelen W, de Haan A. Voluntary activation level and muscle fiber recruitment of human quadriceps during lengthening contractions. J Appl Physiol (1985). 2004 Aug;97(2):619-26. doi: 10.1152/japplphysiol.01202.2003. Epub 2004 Apr 9. PMID 15075302
- [Background] Fitzgerald GK, Piva SR, Irrgang JJ, Bouzubar F, Starz TW. Quadriceps activation failure as a moderator of the relationship between quadriceps strength and physical function in individuals with knee osteoarthritis. Arthritis Rheum. 2004 Feb 15;51(1):40-8. doi: 10.1002/art.20084. PMID 14872454
- [Background] Zarkou A, Stackhouse S, Binder-Macleod SA, Lee SCK. Comparison of techniques to determine human skeletal muscle voluntary activation. J Electromyogr Kinesiol. 2017 Oct;36:8-15. doi: 10.1016/j.jelekin.2017.05.011. Epub 2017 Jun 8. PMID 28649011
- [Background] Wilder MR, Cannon J. Effect of age on muscle activation and twitch properties during static and dynamic actions. Muscle Nerve. 2009 May;39(5):683-91. doi: 10.1002/mus.21233. PMID 19229967
- [Background] Newham DJ, Hsiao SF. Knee muscle isometric strength, voluntary activation and antagonist co-contraction in the first six months after stroke. Disabil Rehabil. 2001 Jun 15;23(9):379-86. doi: 10.1080/0963828001006656. PMID 11394588